CLINICAL TRIAL: NCT06827717
Title: Single-center, Single-arm, Phase II Study of Irinotecan Liposome (II) Combined With Temozolomide and Fluzoparib in the Treatment of Recurrent or Metastatic Ewing Sarcoma
Brief Title: Phase II Study of Irinotecan Liposome (II) Combined With Temozolomide and Fluzoparib in Recurrent or Metastatic Ewing Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jin Wang,MD, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-859-01
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Ewing Sarcoma
Keywords: Ewing sarcoma; irinotecan liposome; temozolomide; fluzoparib; PARP
MeSH Terms: conditions — Sarcoma, Ewing | interventions — irinotecan sucrosofate; Temozolomide; fluzoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- irinotecan liposome (II) + temozolomide + fluzoparib (Experimental): irinotecan liposome (II) combined with temozolomide and fluzoparib
  Interventions: Drug: irinotecan liposome (II) + temozolomide + fluzoparib

INTERVENTIONS:
Drug: irinotecan liposome (II) + temozolomide + fluzoparib — Drug Irinotecan Hydrochloride Liposome Injection（II）56.5mg/m2, IV infusion administered on day 1 of every 28-day cycle until disease progression, unacceptable toxicity or death. Other names: HR070803.
  Drug Fluzoparib 50mg PO bid, administered continuously until disease progression, unacceptable toxicity or death. 28 days as a treatment cycle. Other names: SHR-3162.
  Drug Temozolomide 30mg/m2 PO qd, administered on day 1 to day 5 of every 28-day cycle until disease progression, unacceptable toxicity or death.

SUMMARY:
The current study is an investigator-initiated, single-arm phase 2 study that enrolled patients with recurrent and/or metastatic Ewing sarcoma for the treatment of Irinotecan Liposome (II) Combined with Temozolomide and Fluzoparib as the second-line treatment.

DETAILED DESCRIPTION:
This study is a single-center, single-arm, phase II study evaluating the efficacy and safety of irinotecan liposome (II) combined with temozolomide and fluzoparib in the treatment of recurrent or metastatic ewing sarcoma which progressed on 1st line chemotherapy. Eligible patients will be included in this study and treated according to the protocol. Study treatment will be continued until disease progression, unacceptable toxicity, or patient's decision/consent withdrawal. Local investigators will determine disease progression, radiologic or clinical deterioration. A Simon Two-Stage design will enroll approximately 13 patients into Stage 1, and if criteria are met to move to Stage 2, an additional 16 patients will be enrolled.

PRIMARY OBJECTIVE:

I. To assess the antineoplastic efficacy of irinotecan liposome (II) combined with temozolomide and fluzoparib in the treatment of recurrent or metastatic Ewing sarcoma, as measured by the objective response rate (ORR).

SECONDARY EFFICACY OBJECTIVES:

I. To determine the disease control rate (DCR) for irinotecan liposome (II) combined with temozolomide and fluzoparib in the treatment of recurrent or metastatic Ewing sarcoma.

II. To calculate the duration of response (DOR) for irinotecan liposome (II) combined with temozolomide and fluzoparib in the treatment of recurrent or metastatic Ewing sarcoma.

III. To measure median progression-free survival (PFS) in recurrent or metastatic Ewing sarcoma patients who have received irinotecan liposome (II) combined with temozolomide and fluzoparib.

VI. To measure median overall survival (OS) in recurrent or metastatic Ewing sarcoma patients who have received irinotecan liposome (II) combined with temozolomide and fluzoparib.

SECONDARY SAFETY OBJECTIVE:

I. To assess the toxicity profile of irinotecan liposome (II) combined with temozolomide and fluzoparib in the treatment of recurrent or metastatic Ewing sarcoma according to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.

Exploratory OBJECTIVE:

I. To explore the relationship between mutations and expression of DNA Homologous Recombination Repair (HRR) related genes (such as BRCA1/2, PALB2, etc.) and clinical efficacy (such as ORR, DoR, etc.), as well as resistance mechanisms.

ELIGIBILITY:
Inclusion Criteria:

-1. Patients aged 18 to 75 years (calculated as of the date of signing the informed consent), regardless of gender.

2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2. 3. Histologically confirmed advanced or metastatic Ewing sarcoma, with at least one measurable lesion that has not been treated locally (according to RECIST v1.1, this measurable lesion must have a maximum diameter of ≥ 10 mm on spiral CT scans or a short diameter of ≥ 15 mm for enlarged lymph nodes).

4. The primary tumor or locally recurrent tumor cannot be completely resected through surgery or other local treatments (e.g., stereotactic radiosurgery, argon-helium knife, ultrasound-guided focused ultrasound, etc.); first-line chemotherapy (VAC/IE) has failed, leading to distant metastasis, and the metastatic tumors cannot be completely resected through surgery or other local treatments; or the patient refuses surgery or other local treatments.

5. Expected survival of ≥ 12 weeks. 6. Basic normal function of major organs, with severe abnormalities in blood, heart, lung, liver, kidney, bone marrow functions, or immune deficiency diseases meeting protocol requirements:

1. Complete Blood Count (CBC): (No blood transfusion, use of Granulocyte-Colony Stimulating Factor [G-CSF], or corrective therapy within 14 days prior to screening)

   - Hemoglobin ≥ 90 g/L;
   * Neutrophil count ≥ 1.5 × 10^9/L;
   * Platelet count ≥ 75 × 10^9/L;
2. Biochemical Tests: (No albumin infusion within 14 days)

   * Albumin ≥ 29 g/L;
   * Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal (ULN);
   * Total bilirubin (TBIL) ≤ 1.5 times ULN;
   * Creatinine (Cr) ≤ 1.5 times ULN or Cr clearance > 50 mL/min (Cockcroft-Gault formula):
   * Male: Cr clearance = ((140 - age) × weight) / (72 × blood Cr)
   * Female: Cr clearance = ((140 - age) × weight) / (72 × blood Cr) × 0.85
   * Weight in kg; blood Cr in mg/mL;
   * Urinary protein < 2+ (if urinary protein ≥ 2+, a 24-hour urine protein quantification can be performed, with < 1.0 g in 24 hours allowing for inclusion);
3. Coagulation Function: Activated partial thromboplastin time (APTT) and International Normalized Ratio (INR) ≤ 1.5 × ULN (patients on stable doses of anticoagulants like low molecular weight heparin or warfarin, with INR within the expected therapeutic range, can be screened);
4. Thyroid Function: Thyroid-Stimulating Hormone (TSH) ≤ ULN; if abnormal, T3 and T4 levels should be evaluated, with normal levels allowing for inclusion;
5. Echocardiogram: Left ventricular ejection fraction (LVEF) ≥ 60%. 7. Non-surgically sterile or premenopausal female patients must use a medically approved contraceptive method (such as an intrauterine device, contraceptive pills, or condoms) during the study treatment period and for 6 months after the end of study treatment; non-surgically sterile premenopausal females must have a negative serum or urine HCG test within 7 days prior to study enrollment and must not be breastfeeding; male patients with female partners of childbearing potential should use effective contraception during the study and for 6 months after the last dose of fluzoparib, liposomal irinotecan, or temozolomide.

   8. Understanding the study procedures and methods, voluntarily participating in this trial, and signing the informed consent form in writing, with a full understanding of the trial content, process, and potential adverse reactions.

   Exclusion Criteria:
   * 1. Plans to receive any other anti-tumor treatments during this trial. 2. Received radiotherapy for Ewing sarcoma within 4 weeks prior to the first administration of the study drug, or received other investigational drugs or cell therapies.

     3. Presence of intracranial tumor lesions diagnosed by imaging. 4. History of other active malignancies within the past 5 years, or currently having other active malignancies aside from Ewing sarcoma. Curatively treated localized tumors, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, prostate in situ carcinoma, cervical in situ carcinoma, and breast in situ carcinoma, are allowed.

     5. Presence of clinically symptomatic ascites requiring paracentesis or drainage, or having undergone paracentesis within the last 3 months; only those with small amounts of ascites detected by imaging but without clinical symptoms are excluded; uncontrolled or moderate to severe pleural effusion or pericardial effusion; evidence of intraperitoneal free air that cannot be explained by paracentesis or recent surgical procedures.

     6. History of epilepsy, or having experienced diseases that can induce seizures (including transient ischemic attacks, strokes-not just isolated imaging findings of cerebral ischemia without clinical history, or head trauma with loss of consciousness requiring hospitalization) within 12 months prior to the first administration of the study drug.

     7. Previous treatment with PARP inhibitors, irinotecan, temozolomide, including but not limited to fluzoparib.

     8. History of allergic reactions, including severe drug allergies or drug hypersensitivity; known allergies or intolerances to fluzoparib, liposomal irinotecan, temozolomide, or their excipients.

     9. Severe infections (CTCAE grade > 2) occurring within 4 weeks prior to the first administration of the study drug, such as severe pneumonia requiring hospitalization, bacteremia, or infections with complications; baseline chest imaging indicating active pulmonary inflammation, presence of infection symptoms and signs within 2 weeks before the first administration of the study drug, or requiring oral or intravenous antibiotic treatment (excluding prophylactic use of antibiotics).

     10. Cannot discontinue the use of medications that may affect P-glycoprotein (P-gp) during the study period.

     11. Use of strong or moderate inhibitors or inducers of hepatic drug-metabolizing enzyme CYP3A4 within 14 days prior to the first administration of the study drug.

     12. Presence of factors that impair swallowing, chronic diarrhea, bowel obstruction, or other factors affecting drug intake and absorption.

     13. History of myelodysplastic syndromes (MDS) or acute myeloid leukemia (AML), or having had other malignancies within 5 years prior to the first administration of this study (with the exception of completely resolved in situ cancers and malignancies determined by the investigator to have slow progression).

     14. Co-infection with other viral infections (anti-HCV positive, anti-HIV positive, HBsAg positive) or syphilis infection.

     15. History of immune deficiency (including positive human immunodeficiency virus [HIV] test, other acquired or congenital immune deficiencies) or history of organ transplantation.

     16. Known history of abuse of psychotropic substances, alcoholism, or drug abuse.

     17. Any condition judged by the investigator to pose a significant risk to patient safety or to affect the patient's ability to complete the study (such as poorly controlled hypertension, severe diabetes, thyroid disease, and psychiatric disorders) or any other situation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | From Cycle 1 Day 1 (C1D1) to treatment discontinuation for any reason, average of 4 months
  Objective Response Rate(CR+PR), defined as best overall response (complete or partial response) across all assessment time points, determined using RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Disease Control Rate （DCR） | From Cycle 1 Day 1 (C1D1) to treatment discontinuation for any reason, average of 4 months
  Percentage of patients whose BOR is assessed as CR, PR, or Stable Disease (SD)
Duration of Response （DoR） | From first confirmed CR or PR to confirmed PD, average of 4 months
  The time between the date of the radiological evaluation that first confirmed CR or PR and the date of the radiation evaluation that first confirmed Progressive Disease (PD)
Progression Free Survival (PFS) | From Cycle 1 Day 1 (C1D1) to first documented objective PD or death if PD does not occur, average of 4 months
  Time from C1D1 until the date of objective PD (as assessed by RECIST v1.1) or the date of death (by any cause in the absence of disease progression)
Overall Survival (OS) | From Cycle 1 Day 1 (C1D1) to death from any cause, average of 12 months
  Time from C1D1 until the date of death by any cause. Patients who are still alive at the time of the analysis, or who have become lost to follow-up or withdrawn consent will be censored at their last date known to be alive
Incidence of Adverse Events [safety and tolerability] | From Cycle 1 Day 1 (C1D1) to 30 days after the last dose of study treatment
  Adverse events defined according to Common Terminology for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jin Wang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP